CLINICAL TRIAL: NCT07313943
Title: ANALISI DEI LINFOMI CON ASPETTO TIPO-HODGKIN A FENOTIPO ATIPICO PAX5 NEGATIVO
Brief Title: PAX5-NEGATIVE HODGKIN-LIKE LYMPHOMAS: A DIAGNOSTIC CHALLANGE
Acronym: HL PAX5- 2025
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Elena Sabattini, MD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: HL PAX5- 2025
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Hodgkin or Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — tissue Formalin-fixed, paraffin-embedded samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hodgkin lymphoma (HL) is a lymphoma that arises from peripheral B lymphocytes. However, the neoplastic cells, Hodgkin cells and Reed-Sternberg cells, typically lack most B-cell markers, usually preserving the expression of the transcriptional factor PAX5, only phenotypic clue of B-cell origin.

Morphologically similar cells to those diagnostic Hodgkin and Reed-Sternberg cells can also be observed in other lymphocytic proliferations, including Anaplastic Large Cell Lymphoma (ALCL), which originates from T lymphocytes and which share many features with HL, like strong CD30 expression and usually loss of T-cell markers. However, their clinical course is dramatically different with curability rates of >90% for classical HL and an unfavorable prognosis for ALCL.

PAX5 expression in HL and cytotoxic molecules expression in ALCL tumor cells may be a useful aid for diagnosis. However, in some cases the differential diagnosis is difficult owing to absence of these established markers. Furthermore, clonality analyses on classical HL were focused on Ig regions while TCR clonality has not yet been usefully explored.

Studying the TCR clonal status of tumor cells, correlating it with a more comprehensive immunophenotypic profile and investigating the presence or absence of characteristic rearrangements (such as the JAK2 rearrangement, typical of ALCL lymphomas) could help to resolve the immuno-morphological overlap of the two entities and identify a possible repetitive pattern based on morphological, phenotypic and genetic characteristics.

To this aim we intend to involve the Pathological Anatomy of Tubinga to increase the number of cases and achieve statistical significance, given the relative rarity of this entity

DETAILED DESCRIPTION:
Hodgkin lymphoma (HL) is a lymphoma that originates from peripheral B lymphocytes. However, the neoplastic Hodgkin and Reed-Sternberg cells typically lack most B-cell markers, including CD20, CD79a, CD19, Oct2, and BOB1, and retain only the transcription factor regulating B-cell differentiation, BSAP, encoded by the PAX5 gene. This antigen is generally expressed at a weaker intensity compared to that observed in small reactive B lymphocytes, which serve as internal controls ensuring adequate staining. Moreover, not all neoplastic cells show positivity for PAX5. For this reason, PAX5 immunoreactivity represents the only phenotypic clue to the B-cell origin of classical Hodgkin lymphomas.

The diagnosis of HL is relatively straightforward when this phenotype is present and coexists with other immunomorphological features such as CD30 and CD15 positivity and negativity for B- and T-cell lineage markers, cytotoxic markers, and EMA.

Morphologically similar Hodgkin and Reed-Sternberg-like cells can also be observed in other lymphoid proliferations, including anaplastic large cell lymphoma (ALCL), a lymphoma that also shares with HL a strong expression of CD30.³ ALCL originates from T lymphocytes but, similarly to HL, is highly defective in lineage-specific marker expression, often lacking T-cell markers or expressing only a subset of them. As a cytotoxic T-cell lymphoma, it frequently expresses perforin and typically shows aberrant expression of an epithelial antigen (EMA). Two genetic variants of ALCL exist: one carrying a translocation involving the ALK gene, detectable in tissue by immunohistochemistry, and the ALK-negative variant, which is considerably more challenging to diagnose. Further contributing to diagnostic complexity, ALCL may exhibit architectural patterns and morphology resembling those of HL, to the extent that the WHO classification recognizes a morphological "Hodgkin-like" subtype within ALK-positive ALCL.

In diagnostic practice, rare cases are encountered that morphologically resemble classical HL but are PAX5-negative; these cases may coexpress T-cell markers such as CD3 or CD8, cytotoxic markers (e.g., perforin), and EMA and/or show clonal rearrangement of T-cell receptor genes.⁵ Some reported cases have subsequently developed a true T-cell lymphoma and/or exhibited more frequent relapses, resembling HL cases with poorer prognosis. In some of these cases, rearrangement of the JAK2 gene has been described, a genetic alteration more typically associated with ALCL.

Given the potential immunomorphological overlap between PAX5-negative HL and ALK-negative ALCL, we aim to collect these rare cases to assess whether a recurring pattern of morphological, phenotypic, and genetic features can be identified, based on the data used to establish the diagnosis.

The study is observational, multicenter, international, prospective and retrospective

ELIGIBILITY:
Inclusion Criteria:

* Patients with lymphoma diagnosed as classic Hodgkin's lymphoma with a negative PAX5 marker
* Patients with uncertain differential diagnosis between classical Hodgkin's lymphoma with atypical phenotype (PAX5 negative) and ALK-negative anaplastic large T-cell lymphoma (PAX5 negative)
* Adult males and females at diagnosis
* Availability of the molecular and/or cytogenetic data.

Exclusion Criteria:

* Patients with a diagnosis other than that under study, for whom clinical/histological/molecular information is not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to enroll patients who have referred for diagnosis, from January 2014 to March 2025, at the following hospitals: 1) SSD of Hemolymphopathology IRCCS - Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola-Malpighi and 2) the Pathological Anatomy of Tübingen, Germany
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Atypical Hodgkin Lymphoma | 6/12/24 months
  To identify a characteristic morphological, phenotypic, and genetic pattern for lymphoma cases with an atypical Hodgkin lymphoma and to determine whether there are areas of overlap with ALK-negative anaplastic large cell lymphoma.

SECONDARY OUTCOMES:
Clinical-pathological correlations | 6/12/24 months
  To perform clinical-pathological correlations (OS, PFS, possible therapy and response to therapy)

CONTACTS AND LOCATIONS:
Locations (2):
- Universitätsklinikum Tübingen Institut für Pathologie, Tübingen, Germany
- Irccs Azienda Ospedaliero-Universitaria Di Bologna, Bologna, Italy